CLINICAL TRIAL: NCT05056675
Title: The PENG Block in Elective Hip Surgery and Its Effect on Postoperative Pain and Length of Stay: A Multidisciplinary Prospective Randomized Double-blind Controlled Trial.
Brief Title: The PENG Block in Elective Hip Surgery and Its Effect on Postoperative Pain and Length of Stay.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hôpital Fribourgeois (Other)
Responsible Party: Principal Investigator, Matthieu Hanauer, Attending surgeon, M.D., Hôpital Fribourgeois
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2021-01792
Record Dates: First submitted 2021-08-28; First posted 2021-09-24 (Actual); Last update posted 2024-02-02 (Actual); Status verified 2024-01

CONDITIONS: Pain, Postoperative
Keywords: PENG block; Postoperative pain; Elective hip surgery; Total hip arthroplasty; Surgical hip dislocation
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Intervention Model Description: Interdisciplinary, prospective, double-blind (participant and investigator), placebo-controlled, parallel-group study (experimental study, level of evidence I).
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PENG block for anterior total hip arthroplasty or surgical hip dislocation (Experimental): All patients will undergo the same preoperative, standardized protocol. Upon arrival to the operating theatre, routine, standard pre-medication will be applied before induction of general anesthesia. After intubation, the PENG block is performed. Under sonographic guidance, 20 mL of 0.5% ropivacaine iv is injected.
  Interventions: Procedure: PENG block
- Placebo for anterior total hip arthroplasty or surgical hip dislocation (Placebo Comparator): All patients will undergo the same preoperative, standardized protocol. Upon arrival to the operating theatre, routine, standard pre-medication will be applied before induction of general anesthesia. After intubation, the PENG block is performed. Under sonographic guidance, 20 mL of NaCL 0.9% is injected.
  Interventions: Procedure: Placebo

INTERVENTIONS:
Procedure: PENG block — All patients will undergo the same preoperative, standardized protocol. Upon arrival to the operating room, patients will be placed in supine position. Routine, standard pre-medication will be applied before induction of general anesthesia. After intubation, the PENG block is performed. Under sonographic guidance using a curvilinear probe, puncture will be performed in a lateromedial direction until the needle tip reaches the plane between the iliopsoas tendon and periosteum and between the anterior inferior iliac spine and iliopubic eminence. After a negative aspiration test, the blinded test item will be injected in the plane beneath the iliopsoas muscle. Patients will be randomly assigned to receive the test item (20 mL of ropivacaine 0.5%, Naropin). The anesthesiologist and the surgeon are blinded to the product injected.
  Arms: PENG block for anterior total hip arthroplasty or surgical hip dislocation
Procedure: Placebo — ll patients will undergo the same preoperative, standardized protocol. Upon arrival to the operating room, patients will be placed in supine position. Routine, standard pre-medication will be applied before induction of general anesthesia. After intubation, the PENG block is performed. Under sonographic guidance using a curvilinear probe, puncture will be performed in a lateromedial direction until the needle tip reaches the plane between the iliopsoas tendon and periosteum and between the anterior inferior iliac spine and iliopubic eminence. After a negative aspiration test, the blinded test item will be injected in the plane beneath the iliopsoas muscle. Patients will be randomly assigned to receive the placebo (20 mL of NaCL 0.9%). The anesthesiologist and the surgeon are blinded to the product injected.
  Arms: Placebo for anterior total hip arthroplasty or surgical hip dislocation

SUMMARY:
Effective postoperative pain management in elective hip surgery is crucial for the patients well-being, rapid mobilisation and potential reduction of length of stay. In addition to standard intravenous pain medication, anaesthetic blocks are reportedly effective. Recently, the PENG block, a pericapsular pain block without impairment of the motor function has been introduced in literature and performed at the investigator's hospital (HFR Fribourg, Switzerland) for total hip arthroplasty and surgical hip dislocation - the two most commonly performed elective hip surgeries.

As high-quality evidence on the effectiveness of this novel block is lacking, the investigator's objective is to evaluate the effectiveness of (1) patient-reported pain reduction, (2) total consumption of postoperative morphine, and the length of stay at the hospital.

DETAILED DESCRIPTION:
Forty patients undergoing total hip arthroplasty and 40 patients undergoing surgical hip dislocation will be enrolled in a prospective, double-blind, controlled trial performed at the investigator's hospital.

This study will be the first prospective study evaluating the potential of this pain block in elective hip surgery potentially affecting both patients' postoperative well-being and optimizing costs of the hospital by reducing length of stay.

ELIGIBILITY:
Inclusion Criteria:

* Anterior total hip arthroplasty for hip osteoarthritis
* Surgical hip dislocation for femoro-acetabular impingement (type cam-/pincer)
* Age 16-85 years
* American Society of Anesthesiologists (ASA) physical status 1 to 3

Exclusion Criteria:

* Patient refusal/no informed consent
* Inability to give informed consent
* Lateral approach for total hip arthroplasty
* Bilateral procedure
* Additional osteotomies of the femur and/or acetabulum
* Previous hip & pelvis surgery
* Chronic opioid users
* Known allergy or intolerance to medications used in the trial (local anesthetic, opioid)
* Infection at the injection site
* Body mass index > 40kg/m2
* Spinal anesthesia

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 151 (Actual)
Dates: Start 2022-06-01 (Actual); Primary Completion 2023-04-01 (Actual); Study Completion 2023-11-30 (Actual)

PRIMARY OUTCOMES:
Visual analogue scale (VAS) | Reduction of postoperative pain in the first 24 hours after surgery
  Using a ruler, the score is determined by measuring the distance (cm) on the 10-cm line between the "no pain" anchor and the patient's mark, providing a range of scores from 0 to 10. A higher score indicates greater pain intensity

SECONDARY OUTCOMES:
Total morphine consumption (morphine equivalent dose) | Total consumption of postoperative morphine in the first 24 hours after surgery
  Total morphine consumption in morphine equivalent dose (MED) in the fist 24 hours after surgery.
Length of stay (days) | Length of stay at the hospital (in days) from the day of the surgery (day 0) to the day of discharge, up to a maximum of 7 postoperative days
  The length of hospital stay is measured in days, from the day of surgery (day 0) to the patient's discharge from the hospital. Discharge occurs up to a maximum of 7 days after surgery when the 3 following criteria are met: the scar must be dry, the pain must no longer require morphine and the patient must be able to walk with crutches

CONTACTS AND LOCATIONS:
Overall Officials: Matthieu Hanauer, M.D., Principal Investigator — HFR Fribourg - Hôpital cantonal
Locations (1):
- HFR Fribourg - Hôpital cantonal, Fribourg, Switzerland

IPD SHARING:
Plan to Share IPD: Yes
The IPD and results of this study will be presented at national and international orthopedic meetings and will be submitted to highly-ranked peer reviewed orthopedic journals.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: The study will start in June 2022 and summary data will be published.
Access Criteria: Publication in progress

REFERENCES:
- [Background] Learmonth ID, Young C, Rorabeck C. The operation of the century: total hip replacement. Lancet. 2007 Oct 27;370(9597):1508-19. doi: 10.1016/S0140-6736(07)60457-7. PMID 17964352
- [Background] Birnbaum K, Prescher A, Hessler S, Heller KD. The sensory innervation of the hip joint--an anatomical study. Surg Radiol Anat. 1997;19(6):371-5. doi: 10.1007/BF01628504. PMID 9479711
- [Background] Guay J, Parker MJ, Griffiths R, Kopp S. Peripheral nerve blocks for hip fractures. Cochrane Database Syst Rev. 2017 May 11;5(5):CD001159. doi: 10.1002/14651858.CD001159.pub2. PMID 28494088
- [Background] Giron-Arango L, Peng PWH, Chin KJ, Brull R, Perlas A. Pericapsular Nerve Group (PENG) Block for Hip Fracture. Reg Anesth Pain Med. 2018 Nov;43(8):859-863. doi: 10.1097/AAP.0000000000000847. PMID 30063657
- [Background] Cuschieri S. The CONSORT statement. Saudi J Anaesth. 2019 Apr;13(Suppl 1):S27-S30. doi: 10.4103/sja.SJA_559_18. PMID 30930716
- [Background] Pascarella G, Costa F, Del Buono R, Pulitano R, Strumia A, Piliego C, De Quattro E, Cataldo R, Agro FE, Carassiti M; collaborators. Impact of the pericapsular nerve group (PENG) block on postoperative analgesia and functional recovery following total hip arthroplasty: a randomised, observer-masked, controlled trial. Anaesthesia. 2021 Nov;76(11):1492-1498. doi: 10.1111/anae.15536. Epub 2021 Jul 1. PMID 34196965
- [Background] Bell ML, Kenward MG, Fairclough DL, Horton NJ. Differential dropout and bias in randomised controlled trials: when it matters and when it may not. BMJ. 2013 Jan 21;346:e8668. doi: 10.1136/bmj.e8668. PMID 23338004